CLINICAL TRIAL: NCT06230120
Title: A Sham-Controlled, Randomized Trial of Spinal Cord Stimulation for the Treatment of Pain in Chronic Pancreatitis
Brief Title: Spinal Cord Stimulation for the Treatment of Pain in Chronic Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Soren Schou Olesen, Clinical Professor, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-20200077
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pancreatitis; Chronic Pain
Keywords: Pain; Chronic Pancratitis; Pancreatitis; Spinal Cord Stimulation
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain; Pain; Pancreatitis | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Cord Stimulation (Experimental): A stimulation electrode is placed in the epidural space between the T4-T7 spinal levels and connected to an external electrical pulse generator, which is used for stimulation. The stimulus intensity is initially increased in a ramp-like fashion using high-frequency stimulation at 1000 Hz, with pulse widths of 90 microseconds and intensities increasing from 2 to 14 mA to establish the sensation threshold. After establishing the sensation threshold, the 75 % subthreshold of sensation is used as the stimulation intensity during the active stimulation period.
  Interventions: Device: Spinal Cord Stimulation
- Sham (Sham Comparator): For sham treatment, a similar procedure for establishing the sensation threshold is used, and stimulation at the 75 % subthreshold intensity is initiated, but the stimulation device is turned off 30 seconds after the sensation subthreshold is established.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Spinal Cord Stimulation — Stimulation electrode tip (Vectris™ SureScan MRI percutaneous lead, Medtronic Inc, Minneapolis, US)
  External electrical pulse generator (Wireless External Neurostimulator System (WENS), Medtronic)
  Arms: Spinal Cord Stimulation
Device: Sham — Stimulation electrode tip (Vectris™ SureScan MRI percutaneous lead, Medtronic Inc, Minneapolis, US) with external stimulator turned off
  Arms: Sham

SUMMARY:
Chronic pancreatitis leads to severe abdominal pain in up to 70% of patients, and several studies have proposed it has a neuropathic component. Current treatments often fail to provide adequate pain relief, necessitating new innovations for management. Spinal cord stimulation has been proposed to treat severe neuropathic pain refractory to conventional treatment, but sham-controlled trials have not previously been done in patients with visceral pain. This study will test the effect of spinal cord stimulation in chronic pancreatitis patients with insufficient pain relief from standard therapies.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is a condition causing considerable morbidity, with nearly 0.5 million new cases emerging in Europe every year. It is characterized by a fibro-inflammatory process that progressively damages the pancreas. As the disease advances, most patients experience exocrine pancreatic insufficiency and diabetes, but the most debilitating aspect is severe abdominal pain, which affects about 70% of patients. The pain's origins in CP are complex, typically associated with pancreatic inflammation, ductal obstruction, damage to pancreatic nerves due to inflammation and fibrosis, and resulting neuropathy that triggers sensitization in the pain pathways. This may lead to self-perpetuating pain independent of its initial cause.

Current CP pain management involves conventional analgesics, neuromodulators, and specific endoscopic or surgical interventions for selected cases. However, a substantial number of patients still struggle with inadequate pain relief despite these treatments, necessitating innovative approaches to address CP-associated pain effectively.

Spinal cord stimulation (SCS) is a reversible invasive technique that involves stimulating spinal cord neurons and axons using low-voltage electrical current through leads placed in the epidural space behind the spinal cord dorsal columns. The mechanisms through which neurostimulation may alleviate pain and induce neuroplasticity are intricate and impact multiple neuronal and pain pathways. SCS has shown efficacy in managing neuropathic pain. However, there is a lack of sham-controlled research investigating SCS's effect on visceral pain conditions, including CP.

Hypothesizing that SCS, when compared to sham stimulation, can offer clinically significant pain relief and enhance physical functioning and quality of life in CP patients, an investigator-led, randomized, double-blinded, sham-controlled, cross-over study is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis according to the M-ANNHEIM criteria
* Chronic abdominal pain (pain 3=3days per week in at least 3 months)
* Pain insuficiently treated with patients ussual analgesic treatment
* Patients with signs of obstruction of the pancreatic duct due to a stricture or stone have to undergo endoscopic or surgical decompression prior to enrolment

Exclusion Criteria:

* Patients suffering from painful conditions other than chronic pancreatitis that made them unable to distinguish the pain associated with chronic pancreatitis
* Patients with ongoing alcohol abuse and illegal drug dependencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain relief | At baseline and days 7-10 in each stimulation period
  The difference in pain intensity scores between active and sham stimulations measured using a patient pain diary based on a numeric rating scale where a score of "0" indicated no pain and a score of "10" indicated worst pain imaginable. Pain scores are registered daily for one week prior to intervention and during the two periods of active and sham SCS stimulations.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Immediately after the intervention
  The Patient Global Impression of Change assessed after each stimulation period
The modified Brief Pain Inventory short-form (mBPI-sf) | At baseline an immediately after the intervention
  Differences in the pain and functioning composite scores of the modified Brief Pain Inventory short-form between stimulation period (SCS vs sham)
Comprehensive Pain Assessment Tool short-form (COMPAT-sf) | At baseline an immediately after the intervention
  Differences in the Comprehensive Pain Assessment Tool short-form (COMPAT-sf) total score and subscroes between stimulation periods (SCS vs sham)
Quality of life using SF 36 (short form 36 health survey) | At baseline an immediately after the intervention
  Differences in the SF 36 (short form 36 health survey) total score and subscores between stimulation periods (SCS vs sham)
Symptoms of depression and anxiety as documented by the Hospital Anxiety and Depression Scale (HADS) | At baseline an immediately after the intervention
  Differences in the depression and anxiety scores of Symptoms of depression and anxiety as documented by the Hospital Anxiety and Depression Scale (HADS) between stimulation periods (SCS vs sham)

OTHER OUTCOMES:
Quantitative sensory testing: Pressure algometry | At baseline an immediately after the intervention
  Pain detection and tolerance thresholds (kPa)
Quantitative sensory testing: Repetitive pinprick stimulation | At baseline an immediately after the intervention
  Difference in pain scores (VAS) between 1st and 10th stimulus
Quantitative sensory testing: Cold pressor test | At baseline an immediately after the intervention
  Cold pressor endurance time (seconds)
Quantitative sensory testing: Conditioned pain modulation | At baseline an immediately after the intervention
  Relative change in pressure tolerance threshold before and after cold pressor test (%)

CONTACTS AND LOCATIONS:
Overall Officials: Helga A Gulisano, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Gastroenterology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided